CLINICAL TRIAL: NCT02020226
Title: A Cardiac Safety Study of TH-302 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-414
Record Dates: First submitted 2013-11-14; First posted 2013-12-24 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Solid Tumors
Keywords: TH-302; Solid Tumors; QTc; Cardiac; Evofosfamide
MeSH Terms: interventions — TH 302

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TH-302 (Experimental): 480 mg/m2 by IV infusion over 30 minutes on Days 1, 8, and 15 of each 28-day cycle
  Interventions: Drug: TH-302

INTERVENTIONS:
Drug: TH-302 — 480 mg/m2 30 min IV infusion on Days 1, 8, and 15 of a 28 day cycle

SUMMARY:
The Primary objective of this study is:

1. To determine the cardiac safety of TH-302 in patients with advanced solid tumors

The Secondary objectives are:

1. To assess the pharmacokinetics (PK) of TH-302
2. To evaluate whether there is an association between plasma exposure to TH-302 and its active metabolite, Br-IPM, and effects on cardiac repolarization
3. To assess the safety and antitumor activity of TH-302 in patients with advanced solid tumors

DETAILED DESCRIPTION:
This is an open-label study in patients with advanced solid tumors treated with TH-302 to assess safety, pharmacokinetics, and potential effects on cardiac repolarization and antitumor activity in patients with advanced solid tumors.

A dose of 480 mg/m2 of TH 302 will be administered by IV infusion over 30 minutes on Days 1, 8 and 15 of each 28-day cycle. Evaluations of safety, PK, and ECG parameters of cardiac repolarization will be performed on Study Day 1 and Day 2 of Cycle 1.

Cycles will be repeated every 28 days, until toxicity, progressive disease, patient or investigator decision to discontinue treatment, or until a maximum of six treatment cycles. Patients who are clearly benefitting from the treatment based on anti-cancer disease control and tolerability will be able to continue to receive drug past 6 cycles after discussion with the Sponsor. Tumor assessments will be performed after every 2 cycles during treatment.

The rationale for conducting this study is based on (a) prior data demonstrating the clinical benefit in advanced solid tumors as defined by tumor response or stable disease for at least 4 months, (b) tolerability of TH-302 at the proposed dose, and (c) a requirement to perform a dedicated ECG study to address the clinical evaluation of the potential for QT/QTc interval prolongation of TH-302.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients at least 18 years of age
* Advanced solid tumor for which no other higher priority therapies are available
* ECOG performance status of ) to 1
* Measurable or evaluable disease by RECIST 1.1
* Refractory to standard therapy, relapsed after standard therapy, or have no standard therapy that increases survival at least 3 months
* At least 3 weeks from previous cytotoxic chemotherapy or radiation therapy and at least 5 half-lives or 6 weeks, which ever is shorter, after targeted or biologic therapy
* Acceptable renal function defined as serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance ≥ 60mL/min (by Cockcroft Gault formula)
* Acceptable liver function defined as:

  * Bilirubin ≤ 1.5 x upper limit of normal (ULN); does not apply to patients with Gilbert's syndrome
  * AST (SGOT) and ALT (SGPT) ≤ 3.0 x ULN); if liver metastases are present, then ≤ 5 x ULN is allowed
* Adequate bone marrow function (Absolute neutrophil count (ANC) ≥ 1,500 cells/uL; Platelets (PLT) ≥ 100,000 cells/uL)
* Adequate cardiac conduction by ECG without evidence of second- or third-degree atrioventricular block and meeting all of the following ECG criteria:

  * Heart rate 45-100 beats per minute
  * No evidence of second- or third-degree atrioventricular block
  * QRS interval ≤ 110ms
  * QT interval corrected for heart rate by Fridericia's formula (QTcF) ≤ 480ms
  * PR interval ≤ 200ms
  * No arrhythmia interpreted by the study cardiologist to be clinically significant
* Female patients of childbearing age must have a negative serum HCG test unless prior hysterectomy or menopause (defined as age ≥ 55 and twelve consecutive months without menstrual activity). Female patients should not become pregnant or breast-feed while on this study. Sexually active male and female patients should use effective birth control

Exclusion Criteria:

* Receiving QT-prolonging drugs with a risk of causing torsades de pointes (TdP), unless ECG meets inclusion criteria on a stable dose of the drug and with discussion and agreement with the project clinician
* History of risk factors for TdP, including family history of long QT syndrome
* Sustained systolic blood pressure (BP) >140 mm Hg or <90 mm Hg, diastolic BP >100 mm Hg or <60 mm Hg
* Uncontrolled intercurrent illness, including, but not limited to, myocardial infarction within 6 months, unstable symptomatic ischemic heart disease, active uncontrolled infection requiring systemic therapy, or psychiatric illness/social situations that would limit compliance with study requirements
* Major surgery within the 28 days preceding the first dose of study drug
* Newly diagnosed or uncontrolled cancer-related central nervous system disease
* Receiving medications that are moderate or strong inhibitors or inducers of CYP3A4 or that are sensitive substrate or substrates with a narrow therapeutic index of CYP3A4, CYP2D6, or CYP2C9 (see Appendix D)
* Unwillingness or inability to provide written informed consent and comply with the study protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the potential for QT/QTc interval prolongation of TH-302 in patients with solid tumors | 2 years

SECONDARY OUTCOMES:
Evaluate association between plasma exposure to TH-302 and its active metabolite, Br-IPM, and effects on cardiac repolarization | 2 years
Safety and antitumor activity of TH-302 in patients with advanced solid tumors | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lee Cranmer, MD, PhD, Principal Investigator — The University of Arizona Cancer Center
Locations (2):
- United States (2):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Yuma Regional Cancer Center, Yuma, Arizona

REFERENCES:
- See also: Threshold Pharmaceuticals Company Website — http://www.thresholdpharm.com